CLINICAL TRIAL: NCT06550440
Title: The Impact of Family Integrated Care on the Occurrence of Extrauterine Growth Restriction at Discharge in Very Low Birth Weight Infants: a Multicenter, Retrospective Case-control Study
Brief Title: The Impact of Family Integrated Care on Extrauterine Growth Restriction at Discharge in Very Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240712
Record Dates: First submitted 2024-08-06; First posted 2024-08-13 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Very Low Birth Weight Infant
Keywords: very low birth weight infants; family integrated care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the control group: Very low birth weight infants without extrauterine growth restriction at discharge.
  Interventions: Behavioral: family integrated care
- the case group: Very low birth weight infants with extrauterine growth restriction at discharge.
  Interventions: Behavioral: family integrated care

INTERVENTIONS:
Behavioral: family integrated care — Trained NICU nurses give effective education to parents of children, and regard parents as a part of NICU team, so that they can actively provide positive care for babies instead of passive caregivers. Parents mainly participate in nursing care such as bottle feeding, changing diapers, skin contact and so on.

SUMMARY:
To explore the influence of multi-angle factors, including family integrated care, on extrauterine growth restriction at discharge of very low birth weight infants.

DETAILED DESCRIPTION:
To explore the influence of multi-angle factors, including family integrated care, on extrauterine growth restriction at discharge of very low birth weight infants.Very low birth weight infants admitted to 17 neonatal intensive care units in 8 provinces and cities in southeast China from February 2021 to November 2023 were retrospectively included, which were divided into case group and control group according to whether there was extrauterine growth restriction (defined as the weight below the 10th percentile of children of the same age at discharge). The general situation at birth, the length of hospital stay, the incidence of complications during hospital stay, the feeding situation, the length of family participation care and the perinatal situation of the mother were compared between the two groups. The generalized linear mixed model was used to analyze the influencing factors of extrauterine growth retardation at discharge, and the results of influencing factors were visualized by GraphPad Prism 9.0 software.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns admitted to 17 units in 8 provinces from February 2021 to November 2023;
2. Birth weight < 1500 g, gestational age < 32 weeks;
3. admitted in NICU within 24 hours after birth;
4. premature infants without complications (including bronchopulmonary dysplasia, retinopathy of prematurity, necrotizing enterocolitis, intraventricular hemorrhage and late-onset septicemia) at the time of admission.

Exclusion Criteria:

1. death occurred during hospitalization;
2. Incomplete outcome data (lack of EUGR data at discharge).

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: very low birth weight infants
Sampling Method: Non-Probability Sample
Enrollment: 1255 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
total duration of family integrated care | From the day admitted into the NICU until day on discharge，an average of 2 months.
  Trained NICU staffs effectively educate parents as part of the NICU team so that they can proactively provide active care for the baby, rather than passive caregivers. Parents are primarily involved in care such as bottle feeding, diaper changing, skin-to-skin contact and so on.We calculate total duration of family integrated care in hours.

SECONDARY OUTCOMES:
Birth weight | assessed at birth.
  birth weight in grams
Small for gestational age | assessed at birth.
  birth weight<10th percentile of the neonatal growth curve for infants of the same sex and gestational age
Necrotizing enterocolitis | From the day admitted into the NICU until day on discharge, an average of 2 months.
  diagnosed according to the Bella classification
gestational age | assessed at birth.
  gestational age at weeks

OTHER OUTCOMES:
Bronchopulmonary dysplasia | From the day admitted into the NICU until day on discharge，an average of 2 months.
  oxygen is required at 36 weeks of corrected gestational age or at discharge
Retinopathy of prematurity | From the day admitted into the NICU until day on discharge, an average of 2 months.
  diagnosed according to the International Classification of Retinopathy of Prematurity
Intraventricular hemorrhage | From the day admitted into the NICU until day on discharge，an average of 2 months.
  the diagnosis is based on Paplie's classification
Late-onset sepsis | From the day admitted into the NICU until day on discharge, an average of 2 months.
  sepsis occurs >72h after birth

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Hu, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Qiu MF, Zhang Y, Tang YZ, Dou YL, Wang Y, Lyu TC, Fan QL, Ma YL, Li F, Rong H, Tang YF, Gu WW, Chen XC, Liu D, Wang H, Xiao J, Zhang LL, Wang Y, Ye RM, Li D, Li XX, Pang Y, Lin M, Lin M, Xuan Y, Hu XJ; Research Group of Developmental Care for Very Low Birth Weight Infants in China. An investigation into the impact of family integrated care on extrauterine growth restriction at discharge in very low birth weight infants: a multi-centre study. J Glob Health. 2025 Aug 11;15:04168. doi: 10.7189/jogh.15.04168. PMID 40785514